CLINICAL TRIAL: NCT05303987
Title: Trial of Dexmedetomidine Versus Propofol Sedation for Drug-Induced Sleep Endoscopy in Pediatric Obstructive Sleep Apnea
Brief Title: Dexmedetomidine Versus Propofol Sedation for Drug-Induced Sleep Endoscopy in Pediatric Obstructive Sleep Apnea
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erin Kirkham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Erin Kirkham, Assistant Professor of Otolaryngology-Head and Neck Surgery, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HUM00207865; K23HL153897 (NIH)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Drug-Induced Sleep Endoscopy; Propofol; Dexmedetomidine
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A coordinator and anesthesiologist will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propofol sedation (Experimental): 2.5 mg/kg loading dose, then continue at an infusion of 250 mcg/kg/minute.
  Interventions: Drug: Propofol sedation
- Dexmedetomidine sedation (Experimental): 1 mcg/kg loading dose, then continue at an infusion of 1 mcg/kg/hour
  Interventions: Drug: Dexmedetomidine sedation

INTERVENTIONS:
Drug: Propofol sedation — After induction with sevoflurane then Propofol will be initiated.
  If adequate sedation cannot be attained then a ketamine rescue can be given.
  Arms: Propofol sedation
Drug: Dexmedetomidine sedation — After induction with sevoflurane then Dexmedetomidine will be given.
  If adequate sedation cannot be attained then a ketamine rescue can be given.
  Arms: Dexmedetomidine sedation

SUMMARY:
This research study is designed to learn, first, whether two anesthetics have different effects on collapse seen within the upper airway during sleep endoscopy. A second purpose is to learn whether collapse at several levels of the upper airway is associated with obstructive sleep apnea that persists after adenotonsillectomy, the surgery that removes the tonsils and adenoids.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Obstructive sleep apnea (OSA) by the following criteria: Obstructive Apnea Index (OAI) ≥ 1 or Apnea Hypopnea Index (AHI) ≥ 1.5, confirmed on nocturnal, laboratory-based polysomnography within the previous 12 months scored using American Academy of Sleep Medicine pediatric criteria in an accredited sleep lab.
2. Considered to be a surgical candidate for adenotonsillectomy to treat OSA by an board-certified or board-eligible otolaryngologist.
3. Clinical determination by the child's otolaryngologist surgeon that the child would benefit from sleep endoscopy prior to adenotonsillectomy due to one or more reported risk factors for residual sleep apnea after surgery, which may include:

   1. Obese (>95th percentile of body mass index for age)
   2. Severe preoperative OSA (AHI ≥10 events/hour)
   3. Discordance between awake physical exam (eg. small tonsils) and sleep apnea symptoms or severity;
   4. African American race
   5. Age ≥7 years old
4. Male or Female ages 3.00 - 11.99 years of age at the time of consent
5. Parent/guardian ability to understand and willingness to sign a written informed consent..
6. Parent/guardian must understand/read/speak English or Spanish and be able and willing to complete questionnaires.

Exclusion Criteria:

1. Previous adenotonsillectomy or other upper airway surgery (including tracheostomy) with the exception of isolated adenoidectomy if it occurred >18 months prior to recruitment.
2. Major medical diagnosis that may be exacerbated by the study treatment, pose undue risk to the patient, or that may impact interpretation of study results
3. History of allergic reaction to or contraindication to receiving propofol, dexmedetomidine, ketamine or sevoflurane
4. Allergy to eggs, egg products, soybeans or soybean products.
5. Contraindication to receiving general anesthesia

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean obstruction score at the tongue base | During Drug Induced Sleep Endoscopy (DISE) procedure, as judged subsequently by video review by the three raters
  The degree of obstruction is scored on a 4-point scale as 0% (0), <50% (1), 50-99% (2), or 100% (3). Scores from the 3 surgeons will be averaged for use in analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kirkham, MD MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkham EM, Hoi K, Melendez JB, Henderson LM, Leis AM, Puglia MP 2nd, Chervin RD. Propofol versus dexmedetomidine during drug-induced sleep endoscopy (DISE) for pediatric obstructive sleep apnea. Sleep Breath. 2021 Jun;25(2):757-765. doi: 10.1007/s11325-020-02179-x. Epub 2020 Sep 2. PMID 32876805
- [Background] Mahmoud M, Jung D, Salisbury S, McAuliffe J, Gunter J, Patio M, Donnelly LF, Fleck R. Effect of increasing depth of dexmedetomidine and propofol anesthesia on upper airway morphology in children and adolescents with obstructive sleep apnea. J Clin Anesth. 2013 Nov;25(7):529-41. doi: 10.1016/j.jclinane.2013.04.011. Epub 2013 Oct 2. PMID 24096043
- [Background] Kandil A, Subramanyam R, Hossain MM, Ishman S, Shott S, Tewari A, Mahmoud M. Comparison of the combination of dexmedetomidine and ketamine to propofol or propofol/sevoflurane for drug-induced sleep endoscopy in children. Paediatr Anaesth. 2016 Jul;26(7):742-51. doi: 10.1111/pan.12931. Epub 2016 May 23. PMID 27212000